CLINICAL TRIAL: NCT03798626
Title: Phase Ib Study of Gevokizumab in Combination With Standard of Care Anti-cancer Therapies in Patients With Metastatic Colorectal Cancer, Gastroesophageal Cancer and Renal Cell Carcinoma
Brief Title: Gevokizumab With Standard of Care Anti-cancer Therapies for Metastatic Colorectal, Gastroesophageal, and Renal Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVPM087A2101; 2018-003952-19 (EudraCT Number)
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Gastroesophageal Cancer; Renal Cell Carcinoma
Keywords: colorectal cancer; gastroesophageal cancer; renal cell carcinoma; gevokizumab; bevacizumab; modified FOLFOX6; FOLFIRI; ramucirumab; paclitaxel; cabozantinib; CRC; GEC; RCC; VPM087
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Renal Cell | interventions — gevokizumab; Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil; IFL protocol; Irinotecan; Ramucirumab; Paclitaxel; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: 1st line colorectal cancer (Experimental): Treatment for 1st line metastatic colorectal cancer (mCRC) with Gevokizumab, modified FOLFOX6, bevacizumab
  Interventions: Drug: Gevokizumab; Drug: Bevacizumab; Drug: Modified FOLFOX6
- Cohort B: 2nd line colorectal cancer (Experimental): Treatment for 2nd line mCRC with Gevokizumab, FOLFIRI, bevacizumab
  Interventions: Drug: Gevokizumab; Drug: Bevacizumab; Drug: FOLFIRI
- Cohort C: 2nd line gastroesophageal cancer (Experimental): Treatment for 2nd line metastatic gastroesophageal cancer (mGEC) with Gevokizumab, paclitaxel, ramucirumab
  Interventions: Drug: Gevokizumab; Drug: Ramucirumab; Drug: Paclitaxel
- Cohort D: 2nd or 3rd line renal cell carcinoma (Experimental): Treatment for 2nd or 3rd line metastatic renal cell carcinoma (mRCC) with Gevokizumab, cabozantinib
  Interventions: Drug: Gevokizumab; Drug: Cabozantinib

INTERVENTIONS:
Drug: Gevokizumab — 60 mg/mL concentration; administered intravenously (IV)
  Other Names: VPM087
Drug: Bevacizumab — 25 mg/mL concentration; administered IV
  Arms: Cohort A: 1st line colorectal cancer; Cohort B: 2nd line colorectal cancer
Drug: Modified FOLFOX6 — Oxaliplatin [5 mg/mL concentration; administered IV], leucovorin [10 mg/mL concentration; administered IV] (or levoleucovorin [10 mg/mL concentration; administered IV]), and 5-fluorouracil [50 mg/mL concentration; administered IV]
  Other Names: oxaliplatin, leucovorin, 5-fluorouracil
  Arms: Cohort A: 1st line colorectal cancer
Drug: FOLFIRI — Irinotecan [20 mg/mL concentration; administered IV], leucovorin [10 mg/mL concentration; administered IV] (or levoleucovorin [10 mg/mL concentration; administered IV]), and 5-fluorouracil [50 mg/mL concentration; administered IV]
  Other Names: irinotecan, leucovorin, 5-fluorouracil
  Arms: Cohort B: 2nd line colorectal cancer
Drug: Ramucirumab — 10 mg/mL concentration; administered IV
  Arms: Cohort C: 2nd line gastroesophageal cancer
Drug: Paclitaxel — 6 mg/mL concentration; administered IV
  Arms: Cohort C: 2nd line gastroesophageal cancer
Drug: Cabozantinib — 60 mg tablet; administered orally
  Arms: Cohort D: 2nd or 3rd line renal cell carcinoma

SUMMARY:
This study will determine the pharmacodynamically-active dose of gevokizumab and the tolerable dose of gevokizumab in combination with the standard of care anti-cancer therapy in patients with metastatic colorectal cancer, metastatic gastroesophageal cancer and metastatic renal cell carcinoma, and the preliminary efficacy of gevokizumab in combination with the SOC anti-cancer therapy in subjects with mCRC and mGEC.

ELIGIBILITY:
Key Inclusion Criteria:

For All Cohorts:

* Adult ≥ 18 years old.
* Metastatic disease not amenable to potentially curative surgery and with available archival tumor tissue or fresh tumor tissue biopsy.
* Presence of at least 1 measurable lesion assessed by CT and/or MRI according to RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Adequate bone marrow and organ function per defined criteria in the protocol.
* Recovered from acute laboratory and clinical toxicities of prior anti cancer treatment to NCI CTCAE v5.0 grade ≤1 at time of screening, except alopecia and amenorrhea.

For Cohort A:

• First line metastatic colorectal adenocarcinoma.

For Cohort B:

• Second line metastatic colorectal adenocarcinoma that has progressed on prior line of chemotherapy administered for metastatic disease and which must include a fluoropyrimidine and oxaliplatin.

For Cohort C:

• Second line metastatic gastroesophageal adenocarcinoma that has progressed on prior line of chemotherapy administered for metastatic disease, and which must include a platinum agent and fluoropyrimidine doublet.

For Cohort D:

• Second or third line metastatic renal cell carcinoma with a clear cell component and has received one or two lines of treatment for metastatic disease that included an anti angiogenic agent for at least 4 weeks with radiologic progression on that treatment.

For subjects starting from Part 1a in Cohorts A and B:

* Serum hs CRP at screening ≥ 10 mg/L (per central laboratory assessment).
* Not requiring immediate initiation of anti cancer therapy per investigator's best judgement.

For subjects starting from Part 2 in Cohort C:

• Serum hs CRP at screening ≥ 10 mg/L (per central laboratory assessment).

Key Exclusion Criteria:

For All Cohorts:

* Currently receiving any of the prohibited medications or has contraindications as outlined in the 'Contraindications' to SOC regimen components.
* Symptomatic brain metastases or brain metastases that require directed therapy (such as focal radiotherapy or surgery).
* Suspected or proven immunocompromised state, or infections (as defined in the protocol).
* Conditions that have a high risk of clinically significant bleeding after administration of anti VEGF agents.
* Clinically significant, uncontrolled or recent (within last 6 months) cardiovascular disease.

For Cohort D:

* Concomitant medications, herbal supplements, and/or fruits and their juices that are known as strong inhibitors or inducers of CYP3A4/5, and medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
* Impairment of GI function or GI disease that may significantly alter the absorption of cabozantinib.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Part 1a/b (Cohorts A and B): Change in high-sensitivity C-reactive protein (hs-CRP) after first dose of gevokizumab monotherapy | Baseline, Day 15
  Log scale change of hs-CRP at Day 15 from baseline
Part 1b (Safety run-in): Number of dose limiting toxicities (DLTs) [Cohort C and Cohort D] | First 4 weeks of combination treatment
  DLT is defined as an AE or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the beginning of treatment with gevokizumab in combination with the SOC anti-cancer therapies and meets any of the protocol specified criteria.
Part 1b (Safety run-in): Number of DLTs [Cohort A and Cohort B] | First 6 weeks of combination treatment
  DLT is defined as an AE or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the beginning of treatment with gevokizumab in combination with the SOC anti-cancer therapies and meets any of the protocol specified criteria.
Part 2 (Expansion) and Part 1b (Safety run-in): Progression free survival (PFS) rate [Cohort A subjects at RDE level] | At 15 months
  PFS rate is defined as the percentage of participants who have not progressed or died due to any cause within a specified timeframe after study treatment initiation. Progression will be assessed per investigator assessment using RECIST v1.1.
Part 2 (Expansion) and Part 1b (Safety run-in): Progression free survival (PFS) rate [Cohort B subjects at RDE level] | At 9 months
  PFS rate is defined as the percentage of participants who have not progressed or died due to any cause within a specified timeframe after study treatment initiation. Progression will be assessed per investigator assessment using RECIST v1.1.
Part 2 (Expansion) and Part 1b (Safety run-in): Progression free survival (PFS) rate [Cohort C subjects at RDE level] | At 6 months
  PFS rate is defined as the percentage of participants who have not progressed or died due to any cause within a specified timeframe after study treatment initiation. Progression will be assessed per investigator assessment using RECIST v1.1.

SECONDARY OUTCOMES:
Overall response rate (ORR) per investigator assessment using RECIST v1.1 | Up to 5 years
  ORR is defined as the proportion of subjects with best overall response (BOR) of complete response (CR) or partial response (PR), according to RECIST 1.1
Duration of response (DOR) per investigator assessment using RECIST v1.1 | Up to 5 years
  Duration of response is defined as the time from first documented response of CR or PR to date of first documented progression or death due to any cause, according to RECIST 1.1 criteria
Disease Control Rate (DCR) per investigator assessment using RECIST v1.1 | Up to 5 years
  DCR is defined as the proportion of subjects with a BOR of CR, PR, or stable disease (SD), according to RECIST 1.1.
Overall survival (OS) | Up to 5 years
  OS is defined as the time from date of first dose of study treatment to date of death due to any cause.
PFS by baseline hs-CRP category using RECIST 1.1 [Cohort A and B at RDE level] | Up to 5 years
  PFS is defined as the time from the date of first dosing of study drug to the date of the first documented progression or death due to any cause.
PFS for subjects from Part 1b at doses other than RDE level (Cohort A and Cohort B) | Up to 5 years
  PFS is defined as the time from the date of first dosing of study drug to the date of the first documented progression or death due to any cause.
Number of patients with anti-drug antibodies for gevokizumab in the combination regimens | Up to 5 years
  Incidence of immunogenicity for gevokizumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (32):
- United States (3):
  - University of California LA, Los Angeles, California
  - WA Uni School Of Med, St Louis, Missouri
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Leuven
- Canada (2):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Toronto, Ontario
- Novartis Investigative Site, Santiago, Chile
- Novartis Investigative Site, Brno, Czechia
- Germany (3):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Ulm
- Israel (2):
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Japan (5):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sunto Gun, Shizuoka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (4):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Tainan, Taiwan
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Novartis Pharma AG results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18408